CLINICAL TRIAL: NCT07405749
Title: Incidence and Predictive Factors of Elective Procedure-Related Bleeding in Cirrhotic and Non-Cirrhotic Patients With Clinically Significant Portal Hypertension
Brief Title: Cirrhotic and Non-cirrhotic Patients With Clinically Significant Portal Hypertension
Acronym: PREDIBLEED
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 13663
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cirrhosis, Liver; Portal Hypertension; Clinically Significant Portal Hypertension(CSPH); Gastroesophageal Varices
Keywords: Thrombotic events; porto-systemic collaterals
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alterations in conventional coagulation tests in patients with cirrhosis and/or portal hypertension do not reliably predict bleeding risk, as hemostatic balance is complex and often compensated. Many procedure-related bleeding events are driven by non-coagulatory factors, such as portal hypertension or technical aspects of the procedure. Most commonly performed procedures carry a low risk of bleeding even in the presence of elevated INR or thrombocytopenia, and no validated laboratory thresholds support prophylactic correction. Risk assessment should therefore be based on procedural factors, severity of liver disease, and systemic patient conditions, with correction of modifiable risk factors particularly before high-risk elective procedures.

DETAILED DESCRIPTION:
All cirrhotic and non-cirrhotic patients with clinically significant portal hypertension undergoing elective procedures will be followed to assess the occurrence of major bleeding events and other adverse outcomes. Outcomes will include bleeding events, classified according to ISTH criteria as major, clinically relevant non-major, and minor bleeding; venous and arterial thrombotic events, diagnosed using objective methods and classified as symptomatic or incidental in accordance with ISTH recommendations; and liver-related events, including variceal bleeding, ascites, bacterial infections, and hepatic encephalopathy, clinically assessed during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Ability to provide informed consent;
* Specific signs of CSPH (gastroesophageal varices, porto-systemic collaterals, liver stiffness measurement (LSM) > 25 KPa or spleen stiffness measurement (SSM) > 50 KPa);

Exclusion Criteria:

* Age < 18 years;
* Life expectancy < 6 months;
* Patients unable to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include both cirrhotic and non-cirrhotic inpatients and outpatients with CSPH undergoing elective procedures.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Bleeding and Adverse Events in CSPH Patients Undergoing Elective Procedures | 36-48 months
  To prospectively define the incidence of bleeding and other adverse events in patients with clinically significant portal hypertension (CSPH) who undergo elective low and high risk procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Santopaolo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitaro A. Gemelli IRCSS,UOC Medicina Interna e Gastroenterologia,Largo A. Gemelli,, Roma, Italy